CLINICAL TRIAL: NCT02243137
Title: Effects of Combinated Administration of Lysine Acetylsalicylate Versus Prasugrel and Aspirin on Platelet Aggregation in Healthy Volunteers
Brief Title: Study of Platelet Function After Administration of Aspirin Versus Lysine Acetylsalicylate
Acronym: ECCLIPSE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: David Vivas (Other)
Collaborators: St Carlos Hospital, Madrid, Spain (Other)
Responsible Party: Sponsor-Investigator, David Vivas, MD, PhD, Fundacion Investigacion Interhospitalaria Cardiovascular
Organization: Fundacion Investigacion Interhospitalaria Cardiovascular (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2012-ECCLIPSE-01; 2012-001702-20 (EudraCT Number)
Record Dates: First submitted 2013-06-24; First posted 2014-09-17 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Adverse Effect of Antithrombotic Drugs
MeSH Terms: interventions — Aspirin; Prasugrel Hydrochloride; acetylsalicylic acid lysinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- prasugrel and acetylsalicylic (Active Comparator): single dose of prasugrel 60 mg orally and 300 mg acetylsalicylic acid orally
  Interventions: Drug: acetylsalicylic acid; Drug: prasugrel
- lysine acetylsalicylate and prasugrel (Experimental): single dose of prasugrel 60 mg oral and lysine acetylsalicylate 450 mg intravenous
  Interventions: Drug: prasugrel; Drug: lysine acetylsalicylate

INTERVENTIONS:
Drug: acetylsalicylic acid — Administration: one dose of Acetylsalicylic Acid (300mg)
  Other Names: Adiro
  Arms: prasugrel and acetylsalicylic
Drug: prasugrel — Administration: one loading dose (60mg)
  Other Names: Effient
Drug: lysine acetylsalicylate — Administration: one dose (450mg iv)
  Other Names: Inyesprin
  Arms: lysine acetylsalicylate and prasugrel

SUMMARY:
This is a phase I clinical trial in healthy volunteers comparing the effect of lysine acetylsalicylate or aspirin on platelet function.

DETAILED DESCRIPTION:
1. SUMMARY 1.1. Type of trial Phase I clinical trial in healthy volunteers and marketed drugs 1.2. Identification of the promoter (correspondence to) Dr. David Vivas Balcones Cardiology Department Hospital Clínico San Carlos C/Prof Martín Lagos SN 28040 Madrid Phone: +34 91 330 31 49 Fax: +34 913303142 Email: dvivas@secardiologia.es 1.3. Clinical trial title Effect of combined administration of prasugrel and lysine acetylsalicylate intravenously versus prasugrel and aspirin on platelet aggregation in healthy volunteers (ECCLIPSE trial).

1.4. Protocol code Nº EudraCT: 2012-001702-20 Code: 2012-ECCLIPSE-01 Version: V3 Date: 13/04/2012

1.5. Project principal investigator Dr. David Vivas Balcones Cardiology Department Hospital Clínico San Carlos C/Prof Martín Lagos SN 28040 Madrid Phone: +34 91 330 31 49 Fax: +34 913303142 Email: dvivas@secardiologia.es 1.6. Centers Investigators

San Carlos University Hospital (Madrid). Within the following services and researchers are involved:

Cardiology Department Hospital Clínico San Carlos C/Prof Martín Lagos SN 28040 Madrid Teléfono: +34 91 330 31 49 Fax: +34 913303142 Project principal investigator and Promoter: Dr. David Vivas Balcones Co-Investigators: Dr. Agustín Martín, Dr. Isidre Vilacosta, Dr. Iván Núñez-Gil y Dr. Carlos Macaya

Platelet function laboratory Cardiology Department Hospital Clínico San Carlos C/Prof Martín Lagos SN 28040 Madrid Phone: +34 913307260 Fax: +34 913303142 Co-Investigators: Dr. Antonio Fernández-Ortiz, Esther Bernardo y María Aranzazu Ortega Pozzi

Clinical Trials Unit (CEIC) Biomedical Research Foundation Hospital Clínico San Carlos C/ Prof. Martín Lagos S/N 28040 Madrid Phone: + 34 913303793 Fax: +34 913303515 Co-Investigator: Dra. Saioa Alonso

Clinical Research Ethics Committee The Clinical Research Ethics Committee (CEIC) charged with assessing the project will be the CEIC of the San Carlos University Hospital.

1.7. Responsible for Monitoring: MEDITRIALS 1.8. Experimental and control drug • Experimental group: Loading dose (LD) of intravenous lysine acetylsalicylate 450 mg and prasugrel 60 mg orally.

• Control group: Loading dose (LD) of aspirin 300 mg orally and prasugrel 60 mg orally. Being a crossover study, subjects will receive both treatment arms in the two treatment periods with a gap of 15 days (washout period) between the two administrations.

1.9. Study endpoints Primary endpoint To compare the inhibition of platelet aggregation (IPA) at 30 minutes after administration of prasugrel loading dose in association with intravenous lysine acetylsalicylate versus prasugrel plus aspirin.

Secundary endpoints To compare the inhibition of platelet aggregation (IPA) at 0 (baseline), 1, 4 and 24 hours after the administration of both treatment groups.

To compare the inhibition of platelet reactivity (IPR) throughout the time period in both treatment groups.

To evaluate the safety of the treatment administered.

1.10. Study design The ECCLIPSE study is a phase I, randomized, single center, open, two-period crossover trial in each of which subjects receive a single dose of certain drugs in each treatment group.

1.11. Pathology study None. 1.12. Population and sample size The study population will be healthy volunteers (total 30 subjects). This is a pharmacodynamic study, with subsequent extrapolation of findings to patients with acute coronary syndrome 1.13. Duration of treatment In each period of treatment, subjects will received a single dose of drugs determined in each treatment arm and the analysis of the parameters under study will be processed over the next 24 hours. After the two weeks washout period, subjects will receive the other study drug regimen in a single dose and it will take place the analysis within 24 hours of the parameters studied.

1.14. Primary variable Inhibition of platelet aggregation measured by light transmission aggregometry at 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years.
* BMI> 19kg/m2 and <29kg/m2.
* Women of childbearing potential who are committed to use a medically effective contraception during their participation in the study, except hormonal contraceptives.
* Percentage of inhibition of platelet aggregation after stimulation with high basal 20 mM ADP and arachidonic acid 1.5 mM> 70%.
* No clinically significant deviation on physical examination, ECG or laboratory values in laboratory tests.
* Signed informed consent

Exclusion Criteria:

* Smoking
* Drug abuse
* Pregnant or lactating
* Infection with Hepatitis B or C, or HIV
* Known drug allergies
* Family history of blood disorders or coagulation.
* History of disease that alters the absorption, metabolism or excretion of drugs, including jaundice.
* Personal history of bleeding and / or blood dyscrasias (especially hemophilia, hypoprothrombinemia), including vascular malformations reasonable suspicion.
* History of any medically relevant condition
* Background of major surgery in the last 3 months
* Prescription of chronic medication in the 14 days prior to study participation.
* Participation in another study involving the administration of an investigational product in the last 4 months or a product already on the market in the last three months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Inhibition of platelet aggregation | at 30 minutes
  measured by light transmission aggregometry

SECONDARY OUTCOMES:
Inhibition of platelet aggregation | baseline, 1 h, 4 h and 34 h
  measured by light transmission aggregometry
Inhibition of platelet reactivity | baseline, 1 h, 4 h and 34 h
  by the platelet reactivity index (PRI)
Incidence of adverse events | baseline, 30 min, 1 h, 4 h, and 24 h

CONTACTS AND LOCATIONS:
Overall Officials: David Vivas, MD, PhD, Principal Investigator — San Carlos University Hospital, Madrid Spain
Locations (1):
- Hospital Clínico San Carlos, Madrid, Madrid, Spain

REFERENCES:
- [Derived] Vivas D, Martin A, Bernardo E, Ortega-Pozzi MA, Tirado G, Fernandez C, Vilacosta I, Nunez-Gil I, Macaya C, Fernandez-Ortiz A. Impact of Intravenous Lysine Acetylsalicylate Versus Oral Aspirin on Prasugrel-Inhibited Platelets: Results of a Prospective, Randomized, Crossover Study (the ECCLIPSE Trial). Circ Cardiovasc Interv. 2015 May;8(5):e002281. doi: 10.1161/CIRCINTERVENTIONS.114.002281. PMID 25957056